CLINICAL TRIAL: NCT03132675
Title: A Multicenter Phase 2, Open Label Study of Intratumoral Tavokinogene Telseplasmid (Tavo, pIL-12) + Electroporation With Pembrolizumab in Patients With Stage 3/4 Melanoma Who Are Progressing on Either Pembrolizumab or Nivolumab Treatment
Brief Title: Tavo and Pembrolizumab in Patients With Stage III/IV Melanoma Progressing on Either Pembrolizumab or Nivolumab Treatment
Acronym: Keynote-695
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: OncoSec Medical Incorporated (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMS-I103 (KEYNOTE 695); Keynote-695 (Other: Merck & Co); MK3475-695 (Other: Merck & Co)
Record Dates: First submitted 2017-04-24; First posted 2017-04-28 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Stage III/IV Melanoma
Keywords: Melanoma; pIL-12; pembrolizumab; tavokinogene telseplasmid; Keynote 695; IL-12; IL12; plasmid interleukin-12
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Cohort 1A_Locally advanced/metastatic melanoma: pathological diagnosis of unresectable or metastatic melanoma with progression on pembrolizumab or nivolumab, confirmed according to RECIST v1.1. BRAF V600 mutation-positive melanoma could have received standard of care targeted therapy for advanced or metastatic disease (eg, BRAF/MEK inhibitor, alone or in combination) prior to enrolling on this study; however, progression is not required.
  Cohort 1B_Locally advanced/metastatic melanoma: Subjects will be enrolled in order to collect safety data using the GenPulse generator. Eligibility for enrollment will be the same as that for Cohort 1A.
  Cohort 2_Locally advanced/metastatic melanoma with prior exposure to ipilimumab alone or in combination with nivolumab (or other drug(s)/agent(s)): Eligible subjects will be those with pathological diagnosis of unresectable or metastatic melanoma who have been exposed to ipilimumab alone or in combination with nivolumab (or other drug/agent)
Masking Description: Blinded Independent Central Review
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- tavo-EP plus IV pembrolizumab (Experimental): Intratumoral Tavokinogene Telseplasmid (tavo, pIL 12) plus Electroporation (ImmunoPulse) in Combination with Intravenous Pembrolizumab
  Interventions: Biological: tavokinogene telseplasmid; Biological: Pembrolizumab; Device: ImmunoPulse

INTERVENTIONS:
Biological: tavokinogene telseplasmid — Intratumoral tavokinogene telseplasmid (tavo, pIL-12) delivered by electroporation every 6 weeks
  Other Names: pIL-12; tavo-EP
Biological: Pembrolizumab — Intravenous 3 weekly treatments
  Other Names: Keytruda
Device: ImmunoPulse — Device that electroporates the tavokinogene telseplasmid
  Other Names: tavo-EP

SUMMARY:
Keynote 695 is Phase 2 study of intratumoral tavokinogene telseplasmid (tavo; pIL-12) Electroporation (EP) plus IV Pembrolizumab. Eligible patients will be those with pathological diagnosis of unresectable or metastatic melanoma who are progressing or have progressed on either pembrolizumab or nivolumab.

DETAILED DESCRIPTION:
The study will be comprised of a screening period, a treatment period (up to 2 years), a long term follow-up period, and a survival follow-up period.

Eligible subjects will be treated with TAVO-EP to the accessible lesions on days 1, 5, and 8 every 6 weeks and with IV pembrolizumab (200 mg) on Day 1 of each 3-week cycle for up to 18 TAVO-EP cycles and 35 pembrolizumab cycles (from baseline) of continued treatment (approximately 2 years) or until disease progression. As many accessible lesions may be treated, as deemed feasible by the treating physician, as long as the size of each lesion is greater than 0.3 cm × 0.3 cm.

Long-term Follow-up: All subjects will be followed after End of Treatment (EOT) visit for SAEs (through 90 days from last dose of study drug). Subjects who discontinue treatment will enter the long-term follow-up period unless they have started a new anti-cancer therapy (or other local anticancer immunotherapy) or have withdrawn consent for non-survival assessments. They will have scans, photographs, and investigator-assessed disease evaluation per RECIST v1.1 collected every 3 months until disease progression, or the subject receives a new systemic anti-cancer treatment (or other local anticancer immunotherapy).

Survival Follow-up: Once a subject receives a new systemic anti-cancer treatment (or other local anticancer immunotherapy), they will move into survival follow-up. All subjects will be followed for survival and disease status, every 3 months up to a total duration of 5 years, withdrawal of consent, or until Sponsor terminates the study.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for participation in this study, the subject must meet all of the following:

All Cohorts:

1. Pathologically documented unresectable melanoma, American Joint Committee on Cancer (AJCC) version 8, Stage III or IV. Subjects must have histological or cytological confirmed diagnosis of unresectable melanoma with progressive locally advanced or metastatic disease.
2. Subjects must be refractory to anti-PD-1 monoclonal antibodies (mAb) (pembrolizumab or nivolumab either as monotherapy or in combination with other approved checkpoint inhibitors or targeted therapies according to their approved label) and subjects must meet all of the following criteria:

   1. Received treatment of FDA-approved anti-PD1 mAb (dosed per label of the country providing the clinical site) for at least 12 weeks (eg, 4 administrations of q3w 200 mg pembrolizumab or 2 administrations of q6w 400 mg pembrolizumab).
   2. Progressive disease after anti-PD-1 mAb will be defined according to RECIST v1.1. The initial evidence of PD is to be confirmed by a second assessment, no less than 4 weeks from the date of the first documented PD, in the absence of rapid clinical progression. For cases of rapid clinical progression, patients may be allowed to enroll without a confirmatory scan after discussion with the sponsor. (This determination is made by the Investigator; the Sponsor will collect imaging scans for retrospective analysis. Once PD is confirmed, the initial date of PD documentation will be considered the date of disease progression).
   3. Documented disease progression within 12 weeks of the last dose of anti- PD-1 mAb. Subjects who were re-treated with anti-PD-1 mAb and subjects who were on maintenance with anti-PD-1 mAb will be allowed to enter the study as long as there is documented PD within 12 weeks of the last treatment date (with anti-PD-1 mAb).

   Note: anti-PD-1 combination therapy is acceptable as the last prior treatment and may include, anti-PD-1 anti-CTLA4 antibody combination therapy and anti-PD-1 combinations with investigational or injectable therapy.

   Cohort 2:
3. Subjects must have received ipilimumab alone or in combination with nivolumab (or another agent) within approximately 12 months and must meet the following criteria:

   1. Subject received 4 doses of ipilimumab (alone or in combination) or stopped treatment due to treatment-related adverse event, or investigator determined that the risks of further exposure outweigh the benefits.
   2. Subjects with rapid clinical progression after fewer than 4 doses may be allowed after discussion with the sponsor.

   All Cohorts:
4. Resolution/improvement of anti-PD-1 mAb related adverse events (including immune related AEs; irAEs) back to Grade 0-1 and ≤10 mg/day prednisone (or equivalent dose) for irAEs for at least 2 weeks prior to the first dose of study drug:

   1. No history of common toxicity criteria adverse events (CTCAE) Grade 4 irAEs from anti-PD-1 mAb.
   2. No history of CTCAE Grade 3 requiring steroid treatment (>10 mg/day prednisone or equivalent dose) for >12 weeks or CTCAE Grade 2 pneumonitis regardless of steroid treatment. No history of (non-infectious) pneumonitis or interstitial lung disease that required steroids, and no current pneumonitis or interstitial lung disease.
   3. Minimum of 4 weeks (washout period) from the last dose of anti-PD-1 mAb
5. BRAF V600 mutation-positive melanoma could have received standard of care targeted therapy for advanced or metastatic disease (eg, BRAF/MEK inhibitor, alone or in combination) prior to enrolling on this study; however they do not need to have progressed on this treatment.
6. Age ≥ 18 years of age on day of signing informed consent.
7. Has a performance status of 0 or 1 on the ECOG Performance Scale, collected within 7 days of initial treatment.
8. Have measurable disease based on RECIST v1.1, with at least one anatomically distinct lesion. At least one lesion must meet all the following baseline criteria:

   1. Accessible for electroporation;
   2. Must be accurately measured in at least one dimension (longest diameter in the plane of measurement is to be recorded) Note: Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
9. Demonstrate adequate organ function. All screening laboratories should be performed within 10 days of treatment initiation.
10. Women of childbearing potential must have negative pregnancy test (for serum or urine pregnancy test, within 72 hours or 24 hours, respectively, prior to receiving the first study drug administration). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
11. For women of childbearing potential, must be willing to use an adequate method of contraception from the first day of study treatment (or 14 days prior to the initiation of study treatment for oral contraception) and through at least 120 days following last day of study treatment. Acceptable methods include hormonal contraception (oral contraceptives

    - as long as on stable dose, patch, implant, and injection), intrauterine devices, or double barrier methods (eg, vaginal diaphragm/ vaginal sponge plus condom, or condom plus spermicidal jelly), sexual abstinence or a vasectomized partner. Women may be surgically sterile or at least 1-year post-last menstrual period. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

    Note: Spermicide alone is not considered sufficient and will not be accepted
12. Male subjects must be surgically sterile or must agree to use adequate method of contraception when having sex with women of childbearing potential and refrains from sperm donation during the study treatment period and through at least 120 days following the last day of study drug administration.. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
13. Able and willing to provide written informed consent and to follow study instructions.

Exclusion Criteria:

1. Subject has disease that is suitable for local therapy administered with curative intent.
2. Clinically active CNS metastases. Subjects with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study drug.
3. Subject with a diagnosis of uveal or mucosal melanoma.
4. Subject with clinically unstable or uncontrolled secondary malignancy that is progressing, or requires active treatment are excluded. In addition, subjects who have had a secondary malignancy that has resolved within the last 6 months, are also excluded.
5. Subject who had an allogenic tissue/solid organ transplant.
6. Subjects who have had intervening therapy following confirmed progression on anti-PD-1 therapy or anti-PD-1 combination therapy with the exception of BRAF inhibitors or BRAF/MEK inhibitor combinations.

   Note: anti-PD-1 combination therapy is acceptable as the last prior treatment and may include, anti-PD-1 anti-CTLA4 antibody combination therapy and anti-PD-1 combinations with investigational or injectable therapy.
7. Subjects who have received 4 or more lines of prior therapy, may be allowed to enroll after discussion with the Medical Monitor.
8. Subjects with electronic pacemakers or defibrillators.
9. Subjects who have a known history of Human Immunodeficiency Virus (HIV) (HIV1/2 antibodies). HIV-infected subjects with a history of Kaposi sarcoma and/or Multicentric Castleman Disease.
10. Subjects who have a known history of Hepatitis B or C infections or known to be positive for Hepatitis B antigen (HBsAg) or Hepatitis B virus (HBV) DNA or active. Active Hepatitis C. Active Hep C is defined by a known positive Hep C Ab result and known quantitative HCV RNA results greater than the lower limits of detection of the assay
11. Subject has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug. The use of physiologic doses of corticosteroids may be approved after consultation with the Sponsor.
12. Subjects who have received a live-virus or live-attenuated vaccination within 30 days of the first dose of treatment. Note: Administration of killed vaccines are allowed. Seasonal flu and COVID-19 vaccines that do not contain live virus are permitted.
13. Subject has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
14. Subject has a history of (non infectious) pneumonitis or interstitial lung disease that required steroids or has current pneumonitis or interstitial lung disease.
15. Subject has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
16. Subject has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent, excluding thyroid, hypo adrenal, and diabetes if well controlled.

    Note: Subjects with ≤Grade 2 neuropathy or ≤Grade 2 alopecia and hypopigmentation are an exception to this criterion and may qualify for the study.

    Note: Participants with endocrine-related AEs Grade ≤2 requiring treatment or hormone replacement may be eligible if approved by the Sponsor.

    Note: If subject underwent major surgery or radiation therapy of >30 Gy within 2 weeks of enrollment, they must have recovered adequately from the procedure and/or any complications from the intervention prior to starting study combination therapy.
17. Participation in another clinical study of an investigational anti-cancer agent or has used an investigational device within 30 days of screening.

    Note: Subjects participating in an observational or supportive care study are an exception to this criterion and may qualify for the study with Sponsor approval.

    Note: Subjects who have entered the follow up phase of an investigational study may participate as long as it has been 30 days after the last dose of the previous investigational agent.
18. Subject has known psychiatric or substance abuse disorder that would interfere with the subject's ability to cooperate with the requirements of the study.
19. Subjects who are pregnant or breast-feeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Estimated)
Dates: Start 2017-10-03 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | approximately 2 years
  ORR by blinded independent central review (BICR) based on RECIST v1.1

SECONDARY OUTCOMES:
Objective Response rate (ORR) | approximately 2 years
  ORR by investigator assessment based on RECIST v1.1
Duration of Response (DOR) | approximately 2 years
  DOR by Investigator assessment and BICR based on RECIST v1.1
Progression free survival (PFS) | approximately 2 years
  PFS by investigator assessment and BICR based on RECIST v1.1
Immune Progression Free Survival (iPFS) | approximately 2 years
  iPFS by Investigator assessment and BICR based on iRECIST
Immune Overall Response Rate (iORR) | approximately 2 years
  iORR by Investigator assessment and BICR based on iRECIST
Overall survival (OS) | approximately 2 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Bridget O'Keeffe, PhD, Study Director — OncoSec Medical Incorporated
Locations (33):
- United States (23):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Yuma Regional Medical Center, Yuma Cancer Center, Yuma, Arizona
  - University of California, San Diego, La Jolla, California
  - UCSF Medical Center, San Francisco, California
  - University of Colorado Anschutz Medical Campus University of Colorado Cancer Center, Aurora, Colorado
  - University of Miami Sylvester Cancer Center, Miami, Florida
  - UF Health Cancer Center at Orlando Health, Orlando, Florida
  - Moffit Cancer Center, Tampa, Florida
  - Ochsner Cancer Institute, New Orleans, Louisiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Michigan Medicine Melanoma Oncology Clinic - Rogel Cancer Center, Ann Arbor, Michigan
  - Dartmouth Hitchcock Clinic, Lebanon, New Hampshire
  - Atlantic Health System, Morristown, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Health Quest Systems, Inc., Poughkeepsie, New York
  - Duke University, Durham, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Penn State Health Hershey Medical Center, Hershey, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Texas Oncology/Baylor, Dallas, Texas
  - Houston Methodist Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Australia (6):
  - Westmead Hospital, Westmead, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Cavalry Central Districts Hospital, Elizabeth Vale, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - St John of God Hospital, Subiaco, Western Australia
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli, Italy
- University of Zurich, Dermatology Clinic, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
There is a DSMB charter that makes anonymised data available.

REFERENCES:
- [Derived] Jacobs L, Yshii L, Junius S, Geukens N, Liston A, Hollevoet K, Declerck P. Intratumoral DNA-based delivery of checkpoint-inhibiting antibodies and interleukin 12 triggers T cell infiltration and anti-tumor response. Cancer Gene Ther. 2022 Jul;29(7):984-992. doi: 10.1038/s41417-021-00403-8. Epub 2021 Nov 9. PMID 34754076